CLINICAL TRIAL: NCT04746703
Title: New Imaging Tools to Explore Impact of Bariatric Surgery on Pancreatic Lesions: PACHIBA- Bariatric Surg
Acronym: PACHIBA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP201020
Record Dates: First submitted 2021-01-07; First posted 2021-02-10 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Bariatric Surgery
Keywords: bariatric surgery; pancreatic parameters
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: The investigators propose an exploratory study aiming at assessing the impact of surgical bariatric treatment on the improvement of pancreatic lesions detected by MRI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI before and 6 months after bariatric surgery (Experimental): Recruitment of patient with planned bariatric surgery in Louis Mourier Hospital by the nutritionist, during the preoperative day hospitalisation (performed during the multidisciplinary preparation for bariatric surgery) when patients are deemed eligible for bariatric surgery according to HAS (High Authority of Health) criteria.
  Programming of MRI in the month between preoperative visit and surgery. During this exam without injection of contrast agents in the radiology department of Louis Mourier Hospital, additional sequences with specific acquisitions as previously validated in humans will be performed for the study.
  Bariatric surgery will be performed as in usual care in Louis Mourier hospital. The same MRI will be performed in day hospitalization scheduled 6 months after surgery.
  Interventions: Radiation: Magnetic Resonance Imaging

INTERVENTIONS:
Radiation: Magnetic Resonance Imaging — Pancreatic MRI will be performed in severe-obese patients with a planned bariatric surgery, before and 6 months after bariatric surgery.

SUMMARY:
The investigators propose an exploratory study aiming at assessing the impact of surgical bariatric treatment on the improvement of pancreatic lesions detected by MRI.

Pancreatic MRI will be performed in severe-obese patients with a planned bariatric surgery, before and 6 months after bariatric surgery.

To assess the impact of bariatric surgery on pancreatic Magnetic Resonance Imaging (MRI) parameters in severe-obese patients

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 to 65 years) with a planned for bariatric surgery (sleeve gastrectomy) according to HAS criteria
* Patients with severe obesity (BMI≥35)

Exclusion Criteria:

* Patients with problem of alcohol abuse (previous or current)
* Patients with problems of understanding
* Patients with previous acute or chronic pancreatitis
* Patients with contraindication to MRI (active implantable medical devices, pacemaker, claustrophobia …)
* Inability to undergo MRI due to weight excess
* Pregnant or breastfeeding woman
* Absence of free and informed consent
* Non affiliation to a social security regime or CMU (Universal health coverage)
* Patient under AME (State medical aid)
* Patient deprived of freedom, subject under a legal protective measure
* Patients who have already had bariatric surgery

Secondary exclusion criteria :

* Patients who have undergone bariatric surgery other than a sleeve gastrectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-10-27 (Estimated); Study Completion 2023-10-27 (Estimated)

PRIMARY OUTCOMES:
Quantitative MRI parameters | 6 months after inclusion
  Pancreatic fat content
Quantitative MRI parameters | 6 months after inclusion
  diffusion parameters (mm² / s)
Quantitative MRI parameters | 6 months after inclusion
  transverse magnetization relaxation rate (Hz)
Quantitative MRI parameters | 6 months after inclusion
  longitudinal relaxation rate (Hz)
Quantitative MRI parameters | 6 months after inclusion
  visco-elastic parameters by measure of tissue stiffness (kPa)

SECONDARY OUTCOMES:
Metabolic and anthropometric parameters before and after bariatric surgery | 6 months after inclusion
  BMI
Metabolic and anthropometric parameters before and after bariatric surgery | 6 months after inclusion
  % fat mass in impedance
Metabolic and anthropometric parameters before and after bariatric surgery | 6 months after inclusion
  weight loss in percent of preoperative body weight
Metabolic and anthropometric parameters before and after bariatric surgery | 6 months after inclusion
  excess weight loss
Metabolic and anthropometric parameters before and after bariatric surgery | 6 months after inclusion
  blood pressure
Metabolic and anthropometric parameters before and after bariatric surgery | 6 months after inclusion
  HOMA-IR index
lipids parameters | 6 months after inclusion
  total cholesterol, HDL, LDL, triglycerides

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'obésité et de physiologie, Colombes, France

IPD SHARING:
Plan to Share IPD: No